CLINICAL TRIAL: NCT02187198
Title: Buprenorphine Treatment for Prescription Opioid Dependence
Brief Title: Buprenorphine Treatment for Opioid Dependence
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IP0040
Record Dates: First submitted 2014-07-08; First posted 2014-07-10 (Estimated); Results first posted 2023-03-10 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Opioid Dependence
Keywords: Opioid Dependence; Buprenorphine
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine; Naloxone; Buprenorphine, Naloxone Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Buprenorphine low dose (Experimental): Participants in this arm will receive a low dose (less than or equal to 8/2mg) of buprenorphine for 12 weeks.
  Interventions: Drug: Buprenorphine
- Buprenorphine high dose (Experimental): Participants in this arm will receive a high dose (16-24mg) of buprenorphine for 12 weeks.
  Interventions: Drug: Buprenorphine

INTERVENTIONS:
Drug: Buprenorphine
  Other Names: Naloxone; Suboxone; Buprenex; Subutex

SUMMARY:
Buprenorphine/naloxone (BUP/NLX) treatment is effective for the treatment of prescription opioid dependence, previous studies have not determined the optimum dose of BUP/NLX for this patient population. The goal of this study is to determine if there are differences in clinical efficacy of BUP/NLX tablet in low dose range (less than or equal to 8/2mg) vs. high dose range (greater than or equal to 16, range 16-24mg). The main outcomes of interest will be treatment retention, use of opioids, and the use of other drugs of abuse.

DETAILED DESCRIPTION:
This is a randomized, open-label clinical trial with approximately 9 Veteran opioid dependent men and women. Veterans were randomized to one of two treatment groups: low dose range of buprenorphine (<8mg) vs. high dose range of buprenorphine/naloxone (BUP/NLX (<16mg). During induction into buprenorphine, all participants will be started at a dose of 2mg, and this dose will be increased as needed for stabilization of opioid withdrawal symptoms, up to 8mg for the low dose group, and up to 16mg for the high dose group, within a 5 day period. Participants will be seen on a daily basis (excluding weekends) for the initial 5 day induction. At the end of the 12-week study, participants will either be referred to a buprenorphine clinic if they wish to continue this medication, or if they wish to be drug free, will undergo detoxification from buprenorphine for up to a 4-week period. Follow-up visits, scheduled at 1, 3, and 6 months after study completion.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females between the ages of 18 to 65, current dependence on prescription opioids as evidenced by documented prior treatment for opioid dependence, signs of opiate withdrawal as evidenced by a Clinical Opiate Withdrawal Scale score of 7 or greater, self-reported history of opioid dependence, and a positive urine toxicology for opiates;
2. willingness to be detoxified from opioids for buprenorphine maintenance ;
3. for women of childbearing age, a negative pregnancy test at screening with agreement to use adequate contraception to prevent pregnancy, with monthly pregnancy tests obtained during study participation.

Exclusion Criteria:

1. use of heroin for more than 4 days in the past month;
2. lifetime history of opioid dependence due to heroin alone;
3. ever used heroin intravenously;
4. requirement for current ongoing opioid treatment for adequate pain management;
5. current alcohol, benzodiazepine, barbiturate use with physiologic dependence as determined during screening history and physical,
6. serious unstable medical illness including bradycardia or other arrhythmias, major cardiovascular, renal, endocrine, or hepatic disorders for which buprenorphine treatment is contraindicated or which at the determination of the MD is medically dangerous;
7. serious psychiatric illness including psychosis, bipolar disorder with psychosis:
8. or significant current suicidal or homicidal thoughts necessitating a higher level or care;
9. known allergy or intolerance to buprenorphine.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-03; Primary Completion 2022-02-01 (Actual); Study Completion 2023-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Ralevski, Ph.D., Principal Investigator — Yale University
Locations (1):
- VA Connecticut Healthcare System - West Haven Campus, West Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Buprenorphine Low Dose: Participants in this arm will receive a low dose (less than or equal to 8/2mg) of buprenorphine for 12 weeks.
  Buprenorphine
- Buprenorphine High Dose: Participants in this arm will receive a high dose (16-24mg) of buprenorphine for 12 weeks.
  Buprenorphine
Period: Overall Study
Arm/Group | Buprenorphine Low Dose | Buprenorphine High Dose
Started | 5 | 4
Completed | 4 | 3
Not Completed | 1 | 1
Not completed — did not show up for appointment and did not return calls after week 9 | 1 | 0
Not completed — did not show up for appointment and did not return calls after week 11 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Buprenorphine Low Dose | Buprenorphine High Dose | Total
Number analyzed (Participants) | 5 | 4 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.60 (13.07) | 43.25 (16.72) | 40.67 (14.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 3 | 4 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 4 | 4 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Urine Toxicology for Opiate Use
Description: Will be used to document opioid use, a urine toxicology screening will be completed weekly during study participation (12 week study)
Time Frame: Weeks 1-12
Measure: Count of Participants; unit: Participants
Arm/Group | Buprenorphine Low Dose | Buprenorphine High Dose
Number analyzed (Participants) | 5 | 4
Participants
  Negative urine toxicology for opiates | 2 | 4
  One positive urine toxicology for opiates during 12 week study | 2 | 0
  Two positive urine toxicology for opiates during 12 week study | 1 | 0

2. Primary Outcome: Urine Toxicology
Description: Will be used to document cannabinoid use, a urine toxicology screening will be completed weekly during study participation (12 week study)
Time Frame: Weeks 1-12
Measure: Count of Participants; unit: Participants
Arm/Group | Buprenorphine Low Dose | Buprenorphine High Dose
Number analyzed (Participants) | 5 | 4
Participants
  Negative urine toxicology for cannabinoids | 3 | 3
  Less than 6 positive urine toxicology for cannabinoids during 12 week study | 1 | 0
  More than 6 positive urine toxicology for cannabinoids during 12 week study | 1 | 1

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Buprenorphine Low Dose | Buprenorphine High Dose
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/4
Other Adverse Events (participants affected / at risk) | 0/5 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-23): https://cdn.clinicaltrials.gov/large-docs/98/NCT02187198/Prot_SAP_000.pdf